CLINICAL TRIAL: NCT03392428
Title: TheraP: A Randomised Phase 2 Trial of 177Lu-PSMA617 Theranostic Versus Cabazitaxel in Progressive Metastatic Castration Resistant Prostate Cancer (ANZUP Protocol 1603)
Brief Title: A Trial of 177Lu-PSMA617 Theranostic Versus Cabazitaxel in Progressive Metastatic Castration Resistant Prostate Cancer
Acronym: TheraP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: Australian Nuclear Science and Technology Organisation (ANSTO) (Unknown); Endocyte (Industry); Prostate Cancer Foundation of Australia (PCFA) (Unknown); Australasian Radiopharmaceutical Trials network (ARTnet) (Unknown); Movember Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 1603
Record Dates: First submitted 2017-12-11; First posted 2018-01-08 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Cancer of the Prostate; Metastatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Pluvicto; cabazitaxel

STUDY DESIGN:
Intervention Model Description: Open label, randomised, stratified, 2-arm, phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 177Lu-PSMA617 (Experimental): Patients randomised to the 177Lu-PSMA617 arm will receive 6-8.5GBq of 177Lu-PSMA617 by intravenous injection once every 6 weeks until progressive disease, prohibitive toxicity or a maximum of 6 cycles.
  The first dose will be administered at 8.5GBq, reducing by 0.5GBq with every cycle given (i.e. to 6.0GBq on the sixth cycle, if reached). In some patients who have an exceptional response, treatment will be paused but can be re-commenced up to the maximum of 6 cycles upon progression.
  Interventions: Other: 177Lu-PSMA617
- Cabazitaxel (Active Comparator): Patients randomised to the Cabazitaxel arm will receive 20mg/m2 Cabazitaxel by intravenous infusion once every 3 weeks until progressive disease, prohibitive toxicity or a maximum of 10 cycles.
  Patients in this arm will also receive prednisolone 10mg orally per day for the duration of their cabazitaxel treatment.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Other: 177Lu-PSMA617 — Patients randomised to the 177Lu-PSMA617 arm will receive 6-8.5GBq of 177Lu-PSMA617 by intravenous injection once every 6 weeks until progressive disease, prohibitive toxicity or a maximum of 6 cycles.
  The first dose will be administered at 8.5GBq, reducing by 0.5GBq with every cycle given (i.e. to 6.0GBq on the sixth cycle, if reached). In some patients who have an exceptional response, treatment will be paused but can be re-commenced up to the maximum of 6 cycles upon progression.
  Other Names: Lutetium Prostate-specific membrane antigen
  Arms: 177Lu-PSMA617
Drug: Cabazitaxel — Patients randomised to the Cabazitaxel arm will receive 20mg/m2 Cabazitaxel by intravenous infusion once every 3 weeks until progressive disease, prohibitive toxicity or a maximum of 10 cycles.
  Patients in this arm will also receive prednisolone 10mg orally per day for the duration of their cabazitaxel treatment.
  Other Names: Jevtana
  Arms: Cabazitaxel

SUMMARY:
This open label, randomised, stratified, 2-arm, multicentre, phase 2 trial aims to determine the activity and safety of Lu-PSMA vs cabazitaxel in men with progressive metastatic castration resistant prostate cancer

DETAILED DESCRIPTION:
Despite recent advances in the treatment of prostate cancer, metastatic disease remains incurable.

Prostate specific membrane antigen (PSMA) is present in high quantities on the cell surface of prostate cancers, and is also further increased in metastatic hormone refractory carcinomas. PSMA is an attractive target for both imaging and treatment of prostate cancer. PSMA bound to the radioactive substance Gallium68 (GaPSMA) is rapidly being adopted for imaging prostate cancer using positron emission tomography (PET) scanning.

Radionuclide therapy is an approach for the treatment of cancer that uses tumour targeting agents to deliver high doses of radiation to sites of tumours. The PSMA molecule used for PET imaging can also be labelled with Lutetium177 (Lu177), a radioactive substance.

The aim of this study is to determine the activity and safety of LuPSMA radionuclide therapy.

Patients with metastatic prostate cancer who have progressed despite hormonal therapy and chemotherapy, will be randomised to receive either LuPSMA radionuclide therapy (up to a maximum of 6 cycles of therapy) or cabazitaxel chemotherapy (up to a maximum of 10 cycles of therapy).

200 participants will be recruited from sites across Australia.

The study will determine the effects on PSA response rate (primary endpoint), pain response, progression free survival, quality of life, and frequency and severity of adverse events. Correlative outcomes include associations between PET imaging and clinical outcomes, and biomarkers and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 or older with metastatic adenocarcinoma of the prostate defined by:

   * Documented histopathology of prostate adenocarcinoma OR
   * Metastatic disease typical of prostate cancer (i.e. involving bone or pelvic lymph nodes or para-aortic lymph nodes)
2. Castration-resistant prostate cancer (defined as disease progressing despite castration by orchiectomy or ongoing Luteinizing Hormone-Releasing Hormone (LHRH) analog
3. Progressive disease with rising PSA on 3 consecutive measurements, and PSA ≥ 20 ng/mL
4. Target or non-target lesions according to RECIST 1.1
5. Prior treatment with docetaxel
6. Significant PSMA avidity on 68Ga-PSMA PET/CT, defined as a minimum uptake of SUVmax 20 at a site of disease, and SUVmax > 10 at sites of measurable disease ≥10mm (unless subject to factors explaining a lower uptake, e.g. respiratory motion, reconstruction artefact)
7. ECOG Performance status 0 to 2
8. Assessed by a medical oncologist as suitable for chemotherapy with cabazitaxel
9. Adequate renal function:

   • Cr Cl ≥ 40mL/min (Cockcroft-Gault formula)
10. Adequate bone marrow function:

    * Platelets ≥ 100 x10 billion /L
    * Hb ≥ 90g/L (no red blood cell transfusion in last 4 weeks)
    * Neutrophils > 1.5 x10 billion/L
11. Adequate liver function:

    * Bilirubin < 1.5 x upper limit of normal (ULN) (or if bilirubin is between 1.5-2x ULN, must have a normal conjugated bilirubin)
    * AST or ALT ≤ 2.0 x ULN (or ≤ 5.0 x ULN in the presence of liver metastases)
12. Estimated life expectancy > 12 weeks
13. Study treatment both planned and able to start within 21 days of randomisation
14. Willing and able to comply with all study requirements, including all treatments (cabazitaxel or Lu-PSMA); and, the timing and nature of all required assessments
15. Signed, written informed consent

Exclusion Criteria:

1. Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components
2. Site(s) of disease that are FDG positive with minimal PSMA expression defined as FDG intensity > 68Ga-PSMA activity OR 68Ga-PSMA SUVmax < 10
3. Sjogren's syndrome
4. Prior treatment with cabazitaxel or Lu-PSMA
5. Contraindications to the use of corticosteroid treatment
6. Active malignancy other than prostate cancer
7. Concurrent illness, including severe infection that may jeopardise the ability of the participant to undergo the procedures outlined in this protocol with reasonable safety
8. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse
9. Patients who are sexually active and not willing/able to use medically acceptable forms of barrier contraception

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is looking at prostate cancer which only affects males. The prostate gland is a male reproductive organ
Enrollment: 201 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Prostate Specific Antigen response rate (PSA RR) | Through study completion, on average 4 years
  PSA RR defined as the proportion of participants in each group with a PSA reduction of ≥ 50% from baseline.

SECONDARY OUTCOMES:
Pain Response (PPI and Analgesic Score) | Through study completion, on average 4 years
  Pain response rate, defined as:
  * >=2 point reduction in PPI score from baseline with no increase in analgesic score; and/or
  * >=50% decrease in analgesic score with no increase in PPI PPI: McGill-Melzack Present Pain Intensity Scale (PPI) Analgesic score: Using Morphine Equivalent Daily Dose (MEDD)
Objective Tumour Response Rate | Through study completion, on average 4 years
  Objective Tumour Response Rate - defined as the proportion of participants with a confirmed complete response (CR) or partial response (PR) divided by the total number of participants (using RECIST 1.1).
Progression free survival | Through study completion, on average 4 years
  Progression free survival - the time from randomisation to date of PSA progression (blood samples), pain progression (on PPI) or radiographic progression (PCWG3 for bone and RECIST 1.1 for soft tissue), whichever occurs first
PSA progression free survival | Through study completion, on average 4 years
  PSA progression free survival, defined as the time from randomisation to PSA progression, assessed using PCWG3 criteria on blood test results.
Pain progression free survival | Through study completion, on average 4 years
  Pain progression free survival - defined as the time from randomisation to pain progression (>=1 point increase on PPI from nadir and >=25% increase in analgesic score (MEDD) from nadir, OR need for palliative radiotherapy).
Radiographic progression free survival | Through study completion, on average 4 years
  Radiographic progression free survival - defined as the time from randomisation to radiographic progression (assessed using PCWG3 criteria for bone lesions and RECIST 1.1 for soft tissue lesions).
Health-related quality of life | Through study completion, on average 4 years
  Health-related quality of life, assessed using a composite of the EORTC core quality of life questionnaire (QLQ C-30) and the Patient Disease and Treatment Assessment Form (PDF).
Overall survival | Through study completion, on average 4 years
  Overall survival - time from registration to death from any cause or last known follow-up alive.
Frequency and severity of adverse events | From first study dose to 12 weeks after completing study treatment
  Frequency and severity of adverse events (composite), assessed using CTCAE v4.03.

OTHER OUTCOMES:
Tertiary Correlative objectives: Associations between Ga-68 PSMA PET/CT, FDG-PET/CT baseline characteristics, and outcomes | Through study completion, on average 4 years
  Identification of Ga-68 PSMA PET/CT, FDG-PET/CT markers to predict outcomes.
Tertiary Correlative objectives: Associations between clinical outcomes and possible prognostic and/or predictive biomarkers (tissue and circulating) including ctDNA | Through study completion, on average 4 years
  Identification of biomarkers to predict outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hofman, A/Prof, Study Chair — Peter MacCallum Cancer Centre, Melbourne, Australia
Locations (11):
- Australia (11):
  - Liverpool Hospital, Liverpool, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Royal Brisbane and Womens Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Monash Moorabbin Hospital, Moorabbin, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

REFERENCES:
- [Derived] Kwan EM, Ng SWS, Tolmeijer SH, Emmett L, Sandhu S, Buteau JP, Iravani A, Joshua AM, Francis RJ, Subhash V, Lee ST, Scott AM, Martin AJ, Stockler MR, Donnellan G, Annala M, Herberts C, Davis ID, Hofman MS, Azad AA, Wyatt AW; TheraP Investigators and the ANZUP Cancer Trials Group. Lutetium-177-PSMA-617 or cabazitaxel in metastatic prostate cancer: circulating tumor DNA analysis of the randomized phase 2 TheraP trial. Nat Med. 2025 Aug;31(8):2722-2736. doi: 10.1038/s41591-025-03704-9. Epub 2025 May 27. PMID 40425844
- [Derived] Hofman MS, Emmett L, Sandhu S, Iravani A, Buteau JP, Joshua AM, Goh JC, Pattison DA, Tan TH, Kirkwood ID, Ng S, Francis RJ, Gedye C, Rutherford NK, Weickhardt A, Scott AM, Lee ST, Kwan EM, Azad AA, Ramdave S, Redfern AD, Macdonald W, Guminski A, Hsiao E, Chua W, Lin P, Zhang AY, Stockler MR, Williams SG, Martin AJ, Davis ID; TheraP Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group. Overall survival with [177Lu]Lu-PSMA-617 versus cabazitaxel in metastatic castration-resistant prostate cancer (TheraP): secondary outcomes of a randomised, open-label, phase 2 trial. Lancet Oncol. 2024 Jan;25(1):99-107. doi: 10.1016/S1470-2045(23)00529-6. Epub 2023 Nov 30. PMID 38043558
- [Derived] Viljoen B, Hofman MS, Chambers SK, Dunn J, Dhillon HM, Davis ID, Ralph N. Experiences of participants in a clinical trial of a novel radioactive treatment for advanced prostate cancer: A nested, qualitative longitudinal study. PLoS One. 2022 Nov 9;17(11):e0276063. doi: 10.1371/journal.pone.0276063. eCollection 2022. PMID 36350899
- [Derived] Buteau JP, Martin AJ, Emmett L, Iravani A, Sandhu S, Joshua AM, Francis RJ, Zhang AY, Scott AM, Lee ST, Azad AA, McJannett MM, Stockler MR, Williams SG, Davis ID, Hofman MS; TheraP Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group. PSMA and FDG-PET as predictive and prognostic biomarkers in patients given [177Lu]Lu-PSMA-617 versus cabazitaxel for metastatic castration-resistant prostate cancer (TheraP): a biomarker analysis from a randomised, open-label, phase 2 trial. Lancet Oncol. 2022 Nov;23(11):1389-1397. doi: 10.1016/S1470-2045(22)00605-2. Epub 2022 Oct 16. PMID 36261050
- [Derived] Viljoen B, Hofman MS, Chambers SK, Dunn J, Dhillon H, Davis ID, Ralph N. Advanced prostate cancer experimental radioactive treatment-clinical trial decision making: patient experiences. BMJ Support Palliat Care. 2021 Aug 9:bmjspcare-2021-002994. doi: 10.1136/bmjspcare-2021-002994. Online ahead of print. PMID 34373282
- [Derived] Hofman MS, Emmett L, Sandhu S, Iravani A, Joshua AM, Goh JC, Pattison DA, Tan TH, Kirkwood ID, Ng S, Francis RJ, Gedye C, Rutherford NK, Weickhardt A, Scott AM, Lee ST, Kwan EM, Azad AA, Ramdave S, Redfern AD, Macdonald W, Guminski A, Hsiao E, Chua W, Lin P, Zhang AY, McJannett MM, Stockler MR, Violet JA, Williams SG, Martin AJ, Davis ID; TheraP Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group. [177Lu]Lu-PSMA-617 versus cabazitaxel in patients with metastatic castration-resistant prostate cancer (TheraP): a randomised, open-label, phase 2 trial. Lancet. 2021 Feb 27;397(10276):797-804. doi: 10.1016/S0140-6736(21)00237-3. Epub 2021 Feb 11. PMID 33581798
- [Derived] Iravani A, Violet J, Azad A, Hofman MS. Lutetium-177 prostate-specific membrane antigen (PSMA) theranostics: practical nuances and intricacies. Prostate Cancer Prostatic Dis. 2020 Mar;23(1):38-52. doi: 10.1038/s41391-019-0174-x. Epub 2019 Oct 8. PMID 31595044